CLINICAL TRIAL: NCT05054972
Title: Left Renal Vein Division for Juxtarenal Aortic Exposure: Renal Function and Role of the Communicating Lumbar Vein
Brief Title: Left Renal Vein Division for Juxtarenal Aortic Exposure
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Andreas Selberherr, Dr. Andreas Selberherr, PhD, FEBS, Medical University of Vienna
Other Study IDs: ComLum
Record Dates: First submitted 2021-09-19; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Aortic Aneurysm; Juxtarenal Aortic Aneurysm; Renal Function Disorder
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- A: Group of patients in whom the left renal vein was divided for exposure of the aorta.
  Interventions: Procedure: Exclusion of the aortic aneurysm.
- A+: Subgroup of group A in whom a communicating vein to the left ascending lumbar vein was present.
  Interventions: Procedure: Exclusion of the aortic aneurysm.
- A-: Subgroup of group A in whom a communicating vein to the left ascending lumbar vein was not present.
  Interventions: Procedure: Exclusion of the aortic aneurysm.
- B: Group of patients in whom the left renal vein was mobilized but not divided for exposure of the aorta.
  Interventions: Procedure: Exclusion of the aortic aneurysm.

INTERVENTIONS:
Procedure: Exclusion of the aortic aneurysm. — Surgical procedure in which an aortic aneurysm is excluded.

SUMMARY:
Retrospective study on the outcome of the renal function in patients operated because of juxtarenal aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

Only patients who went for a planned operation because of a juxtarenal aortic aneurysm were included in this retrospective analysis.

Exclusion Criteria:

Emergency surgery Rupture Pending rupture

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were treated surgically for a juxtrarenal aortic aneurysm with an open operation.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Renal function after surgery. | 24 months
  The level of creatinine in the blood was measured after surgery at several time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Vascular Surgery, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided